CLINICAL TRIAL: NCT02623075
Title: Influenza Vaccine Responses as a Means of Assessing Immune Competence in Chimeric Kidney/Stem Cell Transplant Recipients
Status: Completed | Type: Observational
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Joseph Leventhal, Professor of Surgery, Organ Transplantation, Northwestern University
Other Study IDs: STU00201741
Record Dates: First submitted 2015-11-19; First posted 2015-12-07 (Estimated); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines; fluarix

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (3):
- Transplant recipients (Chimeric): Adults who have received a kidney/stem cell transplant and have achieved chimerism will receive the IIV4 (influenza vaccine).
  Interventions: Biological: Influenza vaccine
- Transplant recipients (IS): Adults who have received a kidney/stem cell transplant and are currently maintained on standard immunosuppressive therapy will receive the IIV4 (influenza vaccine).
  Interventions: Biological: Influenza vaccine
- Controls: Healthy adults who meet inclusion and exclusion criteria will receive the IIV4 (influenza vaccine).
  Interventions: Biological: Influenza vaccine

INTERVENTIONS:
Biological: Influenza vaccine — Blood samples will be collected at research study visits at 0 and 30 days (+/- 2 days) post-IIV4 (influenza vaccine). Collection will be as follows: 45-50 ml blood at each visit (not to exceed more than three visits over a two month period).
  Other Names: Fluarix

SUMMARY:
Influenza infection in solid organ transplant recipients is associated with increased morbidity and mortality compared to non-transplanted controls, due in part to the effects of immunosuppression which is necessary to prevent rejection of the transplanted organ. However, transplant patients are less likely to produce antibodies when vaccinated and when they do, the peak and duration of antibody responses are reduced compared to healthy controls. There are considerable differences in the magnitude of these responses, reflecting variability in individual responses to the influenza vaccine and to the immunosuppression regimen. The investigators hypothesize that chimeric kidney transplant recipients off of immunosuppression will have post vaccine immune responses that are comparable to age and gender matched healthy controls.

DETAILED DESCRIPTION:
Influenza infection in solid organ transplant recipients is associated with increased morbidity and mortality compared to non-transplanted controls, due in part to the effects of immunosuppression which is necessary to prevent rejection of the transplanted organ. Annual influenza vaccination is the best way to prevent influenza infection and current CDC, AST Infectious Diseases Community of Practice and American Society for Blood and Marrow Transplantation guidelines recommend annual influenza vaccination to all transplant recipients. However, transplant patients are less likely to produce antibodies when vaccinated and when they do, the peak and duration of antibody responses are reduced compared to healthy controls. There are considerable differences in the magnitude of these responses, reflecting variability in individual responses to the influenza vaccine and to the immunosuppression regimen.

Over the past several years, the investigators have conducted a Phase 2 clinical trial of combined kidney and stem cell transplantation that has been successful in achieving transplantation tolerance in a significant number of recipients. A central tenant for transplantation tolerance is a selective loss of immune reactivity to the allograft while preserving immune responses to all other antigens. The investigators hypothesize that chimeric kidney transplant recipients off of immunosuppression will have post vaccine immune responses that are comparable to age and gender matched healthy controls. The proposed studies aim to assess the immune competence in these fully chimeric tolerant recipients, by quantifying their T and B cell responses to the 2015-2016 inactivated influenza vaccine, quadrivalent (IIV4), standard dose and by testing whether the responding T and B cells arise from memory cells of recipient origin.

These studies will allow the investigators to quantify the influenza -specific cellular, humoral, and molecular responses to IIV4 in tolerant vs. matched controls. On days 0 and 30 days post -IIV4, the flu-specific B cell and neutralizing antibody responses, and the flu-specific IFN-gamma T cell response will be quantified. Additionally, the investigators will perform genome-wide gene expression profiling on isolated PBMC on days 0 and 30 post-IIV4 to characterize the blood response at the transcriptome level.

ELIGIBILITY:
Inclusion Criteria:

* Adults who have received either a combined kidney/stem cell transplant and have achieved chimerism or post-transplant recipients who are maintained on standard immunosuppressive therapy. Additionally, healthy controls of either gender ≥ 18 years of age will also be recruited.
* Subjects must be willing and able to receive the IIV4 and provide blood samples at research visits.
* Subjects must be willing and able to read, understand, and be capable of giving informed consent for prospective enrollment.

Exclusion Criteria

* Subjects less than 18 years of age.
* Any condition that, in the opinion of the attending physician, would place the patient at undue risk by participating. Specific conditions include but are not limited to anemia prohibitive of phlebotomy, coagulopathy or inability to receive the IIV4.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: kidney/stem cell transplant recipients
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2016-12-05 (Actual); Study Completion 2023-12 (Actual)

PRIMARY OUTCOMES:
Analysis of Immune Response in Transplant Recipient Blood Assays | 1 year
  To quantify the response to inactivated influenza vaccine, quadrivalent (IIV4), standard dose in up to 15 tolerance (chimeric) recipients compared to 15 matched, healthy controls and 15 matched, kidney transplant recipients on standard immunosuppression

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Leventhal, MD, PhD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University Comprehensive Transplant Center, Chicago, Illinois, United States